CLINICAL TRIAL: NCT02922543
Title: Revlimid 5 mg Capsules Special Use-results Surveillance of Long Term Use
Brief Title: A Safety and Efficacy Study of Revlimid® 5 mg Capsules in Patients With Relapsed or Refractory Multiple Myeloma Who Have Received Long-term Treatment With it Under the Actual Condition of Use
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-Celgene-JP-PMS-001b
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Teratogenicity; Thrombocytopenia and haemorrhage; Neutropenia and infection; Venous thromboembolism; Allergic reactions; Diarrhoea or constipation; Peripheral neuropathy; Cardiac failure; Arrhythmia; Renal failure; Myocardial infarction; Interstitial lung disease; Tumour lysis syndrome
MeSH Terms: conditions — Multiple Myeloma; Teratogenesis; Thrombocytopenia; Hemorrhage; Neutropenia; Infections; Venous Thromboembolism; Hypersensitivity; Diarrhea; Constipation; Peripheral Nervous System Diseases; Heart Failure; Arrhythmias, Cardiac; Renal Insufficiency; Myocardial Infarction; Lung Diseases, Interstitial; Tumor Lysis Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Relapsed or refractory multiple myeloma (MM) patients: Relapsed or refractory MM patients in the special use-results surveillance (all-case surveillance) (hereinafter referred to as the all-case surveillance) who have received Revlimid treatment for at least 7 cycles at institutions cooperating in performing the all-case surveillance and this surveillance.

SUMMARY:
To understand the safety and efficacy of Revlimid® 5 mg Capsules (hereinafter referred to as Revlimid) in patients with "relapsed or refractory multiple myeloma" (hereinafter referred to as "relapsed or refractory MM") who have received long-term treatment with it under the actual condition of use.

1. Planned registration period This period started on the date of initial marketing of Revlimid and will end at the time when the planned number of patients to be enrolled, 300, is reached (estimated to be approximately 1 year and 3 moths).
2. Planned surveillance period This period started on the date of initial marketing of Revlimid and will end 3 years after the last enrolled patient begins receiving Revlimid (estimated to be approximately 4 years and 3 months).

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory MM patients in the special use-results surveillance (all-case surveillance) (hereinafter referred to as the all-case surveillance) who have received Revlimid treatment for at least 7 cycles at institutions cooperating in performing the all-case surveillance and this surveillance.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Relapsed or refractory multiple myeloma (MM) patients in the special use-results surveillance (all-case surveillance) (hereinafter referred to as the all-case surveillance) who have received Revlimid treatment for at least 7 cycles at institutions cooperating in performing the all-case surveillance and this surveillance.
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2011-02-18 (Actual); Primary Completion 2014-10-11 (Actual); Study Completion 2014-10-11 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 3 years
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Shinko Hospital, Kobe, Hyōgo, Japan